CLINICAL TRIAL: NCT04753606
Title: A Placebo-Controlled, Double-Blind, Randomized, Phase 2 Dose-Finding Study to Evaluate the Effect of Obicetrapib as an Adjunct to High-Intensity Statin Therapy
Brief Title: Randomized Study of Obicetrapib as an Adjunct to Statin Therapy
Acronym: ROSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-201
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2021-09

CONDITIONS: Dyslipidemias; High Cholesterol; Hypercholesterolemia
Keywords: obicetrapib; statin; LDL-C; cholesterol; atherosclerosis
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo tablet made to resemble active
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): once-daily placebo
  Interventions: Drug: Obicetrapib
- obicetrapib 5 mg (Experimental): once-daily obicetrapib
  Interventions: Drug: Obicetrapib
- obicetrapib 10 mg (Experimental): once-daily obicetrapib
  Interventions: Drug: Obicetrapib

INTERVENTIONS:
Drug: Obicetrapib — tablets
  Other Names: CETP inhibitor

SUMMARY:
This study will be a placebo-controlled, double-blind, randomized, phase 2 dose-finding study to evaluate the efficacy, safety, and tolerability of obicetrapib as an adjunct to high-intensity statin therapy.

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, randomized, phase 2 dose-finding study to evaluate the efficacy, safety, and tolerability of obicetrapib as an adjunct to high-intensity statin therapy. The screening period for this study will take up to 2-weeks. Afterwards patients will be randomized to placebo, 5 mg obicetrapib or 10 mg obicetrapib for an 8-week treatment period. After the treatment period, patients will continue for a 4-week safety follow-up and a 15-week PK follow-up.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C > 70 mg/dL and TG < 400 mg/dL,
* Treated with a high-intensity statin therapy

Exclusion Criteria:

* BMI > 40 kg/m
* Significant cardiovascular disease
* HbA1c > 10%
* Uncontrolled hypertension
* Active muscle disease
* GFR < 60 ml/min
* Hepatic dysfunction
* Anemia
* History of malignancy
* Alcohol abuse
* Treatment with investigational product
* Treatment with PCSK9
* Clinically significant condition
* Known CETP inhibitor allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Pinnacle Research Group, Anniston, Alabama
  - National Research Institute - Huntington Park, Huntington Park, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Clinical Trials Research, Sacramento, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Progressive Medical Research, Port Orange, Florida
  - IACT Health, Columbus, Georgia
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Oakland Medical Research Center, Troy, Michigan
  - Diabetes and Endocrinology Consultants, P.C., Morehead City, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Summit Research Group, LLC, Munroe Falls, Ohio
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Health Concepts, Rapid City, South Dakota
  - Juno Research, LL, Houston, Texas
  - Manassas Clinical Research Center, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nicholls SJ, Ditmarsch M, Kastelein JJ, Rigby SP, Kling D, Curcio DL, Alp NJ, Davidson MH. Lipid lowering effects of the CETP inhibitor obicetrapib in combination with high-intensity statins: a randomized phase 2 trial. Nat Med. 2022 Aug;28(8):1672-1678. doi: 10.1038/s41591-022-01936-7. Epub 2022 Aug 11. PMID 35953719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 195 participants were screened; out of 195, 120 participants were randomized.
Period: Overall Study
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Started | 40 | 40 | 40
Completed | 39 | 40 | 40
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Population is defined as all participants who received at least one dose of study drug and had a baseline value for LDL-C assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.77) | 61.1 (8.13) | 62.9 (8.48) | 61.8 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 15 | 53
  Male | 19 | 23 | 25 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 6 | 14
  Not Hispanic or Latino | 37 | 35 | 34 | 106
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 10 | 5 | 22
  White | 32 | 30 | 30 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) Values [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline LDL-C is defined as the last measurement prior to the first dose of study drug. LDL-C was calculated using the Friedewald Formula.
  milligrams per deciliter (mg/dL) | 98.6 (31.09) | 99.2 (30.95) | 94.2 (31.14) | 97.33 (31.06)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [Friedewald]
Description: Mean percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group.LDL-C was calculated using the Friedewald equation unless TG
  ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC),
Time Frame: 8-weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 39 | 40
percent change from baseline | -5.48 (23.357) | -37.97 (27.526) | -43.35 (19.369)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -32.96, 95% CI 2-sided [-44.03 to -21.90], Standard Error of Mean 4.943
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -39.18, 95% CI 2-sided [-50.21 to -28.15], Standard Error of Mean 4.927

2. Primary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [Friedewald]
Description: Median Percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. [Friedewald] LDL-C was calculated using the Friedewald equation unless TG ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC),
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 39 | 40
percent change from baseline | 0 [-57.9 to 40.3] | -42.90 [-81.9 to 72.4] | -45.65 [-78.0 to 26.2]
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -32.96, 95% CI 2-sided [-44.03 to -21.90], Standard Error of Mean 4.943
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -39.18, 95% CI 2-sided [-50.21 to -28.15], Standard Error of Mean 4.927

3. Primary Outcome: LS Mean Percent Change Iin Low-Density Lipoprotein Cholesterol (LDL-C) [Friedewald]
Description: LS mean percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. [Friedewald] LDL-C was calculated using the Friedewald equation unless TG ≥400 mg/dL or LDL-C ≤50 mg/dL; if TG ≥400 mg/dL or LDL-C ≤50 mg/dL, then LDL-C level was measured directly by preparative ultracentrifugation (PUC),
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 40 | 40 | 40
percent change from baseline | -5.00 (3.502) | -37.97 (3.491) | -44.18 (3.461)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -32.96, 95% CI 2-sided [-44.03 to -21.90], Standard Error of Mean 4.943
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -39.18, 95% CI 2-sided [-50.21 to -28.15], Standard Error of Mean 4.927

4. Primary Outcome: Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [PUC]
Description: Mean Percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 38 | 40
percent change from baseline | -7.11 (20.773) | -35.98 (25.469) | -46.06 (19.393)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -28.94, 95% CI 2-sided [-38.14 to -19.74], Standard Error of Mean 4.643
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -40.07, 95% CI 2-sided [-49.16 to -30.97], Standard Error of Mean 4.591

5. Primary Outcome: Median Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [PUC]
Description: Median Percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. LDL-C level was measured by preparative ultracentrifugation (PUC).
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 38 | 40
percent change from baseline | -6.50 [-53.9 to 31.6] | -41.45 [-71.2 to 62.3] | -50.75 [-76.9 to 15.6]
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -28.94, 95% CI 2-sided [-38.14 to -19.74], Standard Error of Mean 4.643
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -40.07, 95% CI 2-sided [-49.16 to -30.97], Standard Error of Mean 4.591

6. Primary Outcome: LS Mean Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) [PUC]
Description: LS Mean Percent change from Day 1 to Day 56 in Low-Density Lipoprotein Cholesterol (LDL-C) for each obicetrapib group compared to the placebo group. LDL-C level was measured directly by preparative ultracentrifugation (PUC).
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 38 | 40
percent change from baseline | -6.70 (3.263) | -35.65 (3.305) | -46.77 (3.225)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -28.94, 95% CI 2-sided [-38.14 to -19.74], Standard Error of Mean 4.643
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, ANCOVA; Least Squares (LS) Means = -40.07, 95% CI 2-sided [-49.16 to -30.97], Standard Error of Mean 4.591

7. Secondary Outcome: Mean Percent Change in Apolipoprotein B (ApoB)
Description: Mean percent change from baseline to Day 56 in apolipoprotein B (ApoB) (mg/dL) for each obicetrapib group compared with the placebo group.
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 39 | 40
percent change from baseline | -4.67 (17.687) | -22.62 (21.882) | -27.19 (15.329)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -18.26, 95% CI 2-sided [-25.51 to -11.02], Standard Error of Mean 3.657
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -23.99, 95% CI 2-sided [-31.22 to -16.76], Standard Error of Mean 3.650

8. Secondary Outcome: Median Percent Change in Apolipoprotein B (ApoB)
Description: Median percent change from baseline to Day 56 in apolipoprotein B (ApoB) (mg/dL) for each obicetrapib group compared with the placebo group.
Time Frame: 8-Week
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 39 | 40
percent change from baseline | -2.60 [-50.0 to 28.4] | -24.40 [-58.5 to 47.4] | -29.75 [-58.4 to 13.0]
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -18.26, 95% CI 2-sided [-25.51 to -11.02], Standard Error of Mean 3.657
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -23.99, 95% CI 2-sided [-31.22 to -16.76], Standard Error of Mean 3.650

9. Secondary Outcome: LS Mean Percent Change in Apolipoprotein B (ApoB)
Description: as for outcome 8
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 40 | 40 | 40
percent change from baseline | -4.13 (2.593) | -22.40 (2.582) | -28.12 (2.564)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -18.26, 95% CI 2-sided [-25.51 to -11.02], Standard Error of Mean 3.657
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -23.99, 95% CI 2-sided [-31.22 to -16.76], Standard Error of Mean 3.650

10. Secondary Outcome: Mean Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Mean percent change from baseline to Day 56 in non-high-density lipoprotein cholesterol (non-HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group
Time Frame: 8-weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 39 | 40
percent change from baseline | -4.22 (20.440) | -34.28 (25.623) | -39.25 (17.625)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -30.54, 95% CI 2-sided [-39.46 to -21.62], Standard Error of Mean 4.503
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -36.03, 95% CI 2-sided [-44.92 to -27.14], Standard Error of Mean 4.488

11. Secondary Outcome: Median Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Median percent change from baseline to Day 56 in non-high-density lipoprotein cholesterol (non-HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 39 | 40
percent change from baseline | -3.50 [-50.3 to 48.4] | -38.90 [-65.6 to 66.3] | -44.40 [-70.2 to 22.5]
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -30.54, 95% CI 2-sided [-39.46 to -21.62], Standard Error of Mean 4.503
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -36.03, 95% CI 2-sided [-44.92 to -27.14], Standard Error of Mean 4.488

12. Secondary Outcome: LS Mean Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: LS Mean percent change from baseline to Day 56 in non-high-density lipoprotein cholesterol (non-HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 40 | 40 | 40
percent change from baseline | -3.83 (3.191) | -34.37 (3.179) | -39.86 (3.153)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -30.54, 95% CI 2-sided [-39.46 to -21.62], Standard Error of Mean 4.503
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = -36.03, 95% CI 2-sided [-44.92 to -27.14], Standard Error of Mean 4.488

13. Secondary Outcome: Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C)
Description: Mean percent change from baseline to Day 56 in High-density lipoprotein cholesterol (HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group.
Time Frame: 8-weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 39 | 40
percent change from baseline | -6.62 (12.436) | 123.92 (57.671) | 156.41 (52.165)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 129.27, 95% CI 2-sided [110.78 to 147.77], Standard Error of Mean 9.337
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 164.33, 95% CI 2-sided [145.90 to 182.76], Standard Error of Mean 9.306

14. Secondary Outcome: Median Percent Change in High-density Lipoprotein Cholesterol (HDL-C)
Description: Median percent change from baseline to Day 56 in High-density lipoprotein cholesterol (HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group.
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 39 | 39 | 40
percent change from baseline | -4.90 [-30.3 to 28.6] | 135.40 [-26.4 to 212.9] | 164.95 [55.1 to 286.3]
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 129.27, 95% CI 2-sided [110.78 to 147.77], Standard Error of Mean 9.337
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 164.33, 95% CI 2-sided [145.90 to 182.76], Standard Error of Mean 9.306

15. Secondary Outcome: LS Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C)
Description: LS mean percent change from baseline to Day 56 in High-density lipoprotein cholesterol (HDL-C) (mg/dL) for each obicetrapib group compared with the placebo group.
Time Frame: 8-Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
Number analyzed (Participants) | 40 | 40 | 40
percent change from baseline | -6.98 (6.620) | 122.29 (6.585) | 157.35 (6.538)
Statistical Analysis 1: Comparison: Placebo vs Obicetrapib 5 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 129.27, 95% CI 2-sided [110.78 to 147.77], Standard Error of Mean 9.337
Statistical Analysis 2: Comparison: Placebo vs Obicetrapib 10 mg; Test type: Superiority; p < .0001, Mixed Models Analysis; mixed model for repeated measures (MMRM) with missing at random assumption; Least Squares (LS) Means = 164.33, 95% CI 2-sided [145.90 to 182.76], Standard Error of Mean 9.306

ADVERSE EVENTS:
Time Frame: From first dose of study drug through week 12
Description: Safety Population included all participants who received at least 1 dose of any study drug.
Arm/Group | Placebo | Obicetrapib 5 mg | Obicetrapib 10 mg
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 17/40 | 15/40 | 8/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Obicetrapib 5 mg (N=40) | Obicetrapib 10 mg (N=40)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Obicetrapib 5 mg (N=40) | Obicetrapib 10 mg (N=40)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study, whichever occurs first, Institution may publish the results of its study data. Institution and PI shall provide sponsor with an advance copy of any proposed communications at least 60 days prior and Sponsor shall have 60 days to review. Sponsor may request (a) the deletion of any Confidential Information, (b) reasonable changes, or (c) a delay for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT04753606/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT04753606/SAP_001.pdf